CLINICAL TRIAL: NCT03675373
Title: A Pilot Study on the Feasibility of Alcohol Brief Intervention Plus Personalized Mobile Chat-based Intervention to Reduce High-risk Drinking Among University Students in Hong Kong
Brief Title: Alcohol Brief Intervention Plus Personalized Mobile Chat-based Intervention for High-risk Drinking University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pilot alcohol study (Unists)
Record Dates: First submitted 2018-09-16; First posted 2018-09-18 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Drinking in College
Keywords: chat-based intervention; alcohol brief intervention; high-risk drinking; university students; AUDIT; instant messaging; WhatsApp
MeSH Terms: conditions — Alcohol Drinking in College | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Alcohol brief intervention+mobile chat-based instant messages
  Interventions: Behavioral: Mobile chat-based instant messages; Behavioral: Alcohol brief intervention
- control group (Active Comparator): Alcohol brief intervention
  Interventions: Behavioral: Alcohol brief intervention

INTERVENTIONS:
Behavioral: Mobile chat-based instant messages — Subjects in the active arm study will receive continuous interactive chat-based intervention as an extension of alcohol brief intervention at baseline. The interactive mobile chat will be carried out on Friday night and Saturday before and during the period of "happy hour" and ask for drinking and giving personalized advises on drinking reduction using behavioral change techniques.
  Arms: Intervention group
Behavioral: Alcohol brief intervention — Those in the control arm will be assigned to only receive the face-to-face ABI. The ABI consists of: (1) giving feedback and information about the screening result in phase I and hazard of drinking; (2) emphasizing the benefits of reduce drinking and informing about alcohol problems; (3) setting goal on reducing alcohol consumption; (4) reviewing advice and ;(5) giving encouragement.
  Other Names: ABI

SUMMARY:
The aims of this pilot study are:

1. To examine the factors associated with alcohol drinking and alcohol use disorder
2. To examine the effect of face-to-face alcohol brief intervention on drinking reduction
3. To examine the effect of a continuous interactive chat-based intervention via "WhatsApp" on drinking reduction
4. To explore the perception of face-to-face alcohol brief intervention
5. To explore the perception of continuous interactive chat-based intervention via instant messaging mobile application "WhatsApp"

DETAILED DESCRIPTION:
According to the Department of Health, majority of people in Hong Kong started to develop drinking habit at 18-21 years of age in 2014/2015. Amongst them, 16.8% had scored higher than 3 in the Alcohol Use Disorders Identification Test for Consumption (AUDIT-C) (an abbreviated version of the Alcohol Use Disorders Identification Test, or AUDIT, designed by the World Health Organization(WHO)), while 3.5% had even scored 8 or above in the test. With higher prevalence to begin drinking within 18 and 23 years old, university students could have established higher tendency of harmful drinking and alcohol dependence as compared with other age groups. Therefore, early interventions such as the evidence-based Alcohol Brief Intervention (ABI) suggested by the WHO are particularly needed to target university drinkers who are 5% more likely to develop higher frequency of drinking in later of their lives compared with other age groups.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong resident aged 18 to 26 inclusive
* Scored 5-19 inclusive in the Alcohol Use Disorder Identification Test (AUDIT)
* Able to communicate in Chinese and read Chinese
* Using a phone with instant messaging mobile application "WhatsApp" installed for communication

Exclusion Criteria:

* Students with communication barrier (either physically or cognitively)
* Currently participating in other alcohol treatment services or clinics.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2018-11-04 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in AUDIT score | 2 weeks after baseline
  Assessed by Alcohol Use Disorders Identification Test (ranged 0-40 with higher score indicating problematic alcohol use)

SECONDARY OUTCOMES:
Change in number of standard drinks | 2 weeks after baseline
  Defined by either increase or decrease in standard drinks number
Attempt to reduce drinking | 2 weeks after baseline
  Have tried to reduce drinking either successful or not
Change in confidence to reduce drinking | 2 weeks after baseline
  Defined by either increase or decrease confidence in reduce drinking

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided